CLINICAL TRIAL: NCT05030233
Title: Pilot Study of Nurse-Administered Touch and Biobehavioral Stress Responses of Preterm Infants
Brief Title: Pilot Study of Nursing Touch and Biobehavioral Stress
Acronym: P-NAT-BIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Marliese Nist, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021N0006
Record Dates: First submitted 2021-08-23; First posted 2021-09-01 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Prematurity; Stress Reaction
Keywords: preterm infant; stress; nursing care; touch
MeSH Terms: conditions — Premature Birth; Fractures, Stress

STUDY DESIGN:
Intervention Model Description: randomized cross-over design
Masking Description: The statistician performing the data analysis will be blinded to group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-Administered Touch Intervention (Experimental): Preterm infants will receive the nurse-administered touch intervention during one episode of essential nursing care.
  Interventions: Behavioral: Nurse-Administered Touch Intervention
- Standard Care (No Intervention): Preterm infants will receive one episode of essential nursing care delivered as standard care.

INTERVENTIONS:
Behavioral: Nurse-Administered Touch Intervention — The nurse-administered touch intervention is a bare-handed, comforting touch intervention administered during an episode of essential nursing care. The bedside nurse will cradle the infant's head with one hand, using the other hand to gently support the infant's lower body and legs in a flexed position. The touches will be administered for 1 minute at the start of the essential care episode, 30 seconds after the diaper change, and 1 minute at the conclusion of the care episode.
  Arms: Nurse-Administered Touch Intervention

SUMMARY:
Randomized cross-over clinical trial to determine the effect of a nurse-administered comforting touch intervention on the biobehavioral stress responses of preterm infants hospitalized in the neonatal intensive care unit.

DETAILED DESCRIPTION:
Preterm infants will receive one episode of essential nursing care as standard care and one episode of essential nursing care that includes a nurse-administered comforting touch intervention approximately 24 hours apart in a randomized sequence. For 10 minutes prior to the start of the two observed care episodes, during the care episodes, and for 60 minutes after the conclusion of the care episodes, researchers will measure infants' biobehavioral stress responses. When infants reach 35 weeks post-menstrual age, researchers will perform a neurobehavioral assessment.

ELIGIBILITY:
Inclusion Criteria:

* Born prematurely between 27 and 30 weeks post-menstrual age.
* Born to mothers who are English-speaking and able to provide informed consent.
* No more than 10 days old at the time of enrollment.

Exclusion Criteria:

* Diagnosed with Grade III/IV intraventricular hemorrhage or other neurologic abnormality (e.g. seizure disorder) affecting sensory perception or motor function.
* Diagnosed with a congenital anomaly requiring surgery during the neonatal period.
* Receiving scheduled steroids or vasopressors.
* Skin conditions that preclude the attachment of sensors.
* Diagnosed with Neonatal Abstinence Syndrome or born to mothers with known illicit drug use, except marijuana, during pregnancy.
* Diagnosed with chromosomal abnormalities.
* Requiring special isolation with universal gloving for potentially infectious pathogens.

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marliese D. Nist, PhD, Principal Investigator — Ohio State University
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Nurse-Administered Touch Intervention, Then Standard Care: Preterm infants will receive the nurse-administered touch intervention during one episode of essential nursing care followed by a 24-hour washout period. Then, infants will receive one episode of essential nursing care provided as standard care.
  Nurse-Administered Touch Intervention: The nurse-administered touch intervention is a bare-handed, comforting touch intervention administered during an episode of essential nursing care. The bedside nurse will cradle the infant's head with one hand, using the other hand to gently support the infant's lower body and legs in a flexed position. The touches will be administered for 1 minute at the start of the essential care episode, 30 seconds after the diaper change, and 1 minute at the conclusion of the care episode.
  Standard Care: Essential nursing care includes activities to address infant clinical and hygiene needs and may include discretionary comforting touch. Systematic comforting touch is not routine.
- Experimental: Standard Care, Then Nurse-Administered Touch Intervention: Preterm infants will receive one episode of essential nursing care delivered as standard care followed by a 24-hour washout period. Then, infants will receive one episode of essential nursing care that includes the nurse-administered touch intervention.
  Standard Care: Essential nursing care includes activities to address infant clinical and hygiene needs and may include discretionary comforting touch. Systematic comforting touch is not routine.
  Nurse-Administered Touch Intervention: The nurse-administered touch intervention is a bare-handed, comforting touch intervention administered during an episode of essential nursing care. The bedside nurse will cradle the infant's head with one hand, using the other hand to gently support the infant's lower body and legs in a flexed position. The touches will be administered for 1 minute at the start of the essential care episode, 30 seconds after the diaper change, and 1 minute at the conclusion of the care episode.
Period: Overall Study
Arm/Group | Experimental: Nurse-Administered Touch Intervention, Then Standard Care | Experimental: Standard Care, Then Nurse-Administered Touch Intervention
Started | 10 | 9
Completed | 9 | 9
Not Completed | 1 | 0
Not completed — withdrawn for transfer | 1 | 0

BASELINE CHARACTERISTICS:
Population: 10 infants assigned to receive nurse-administered touch intervention followed by standard care sequence; 9 infants assigned to receive standard care followed by nurse-administered touch intervention sequence
Groups:
- Experimental: Standard Care, Then Nurse-Administered Touch Intervention: Preterm infants will receive one episode of essential nursing care delivered as standard care followed by a 24-hour washout period. Then, infants will receive an episode of essential nursing care that includes the nurse-administered touch intervention.
  Standard Care: Essential nursing care includes activities to address infant clinical and hygiene needs and may include discretionary comforting touch. Systematic comforting touch is not routine.
  Nurse-Administered Touch Intervention: The nurse-administered touch intervention is a bare-handed, comforting touch intervention administered during an episode of essential nursing care. The bedside nurse will cradle the infant's head with one hand, using the other hand to gently support the infant's lower body and legs in a flexed position. The touches will be administered for 1 minute at the start of the essential care episode, 30 seconds after the diaper change, and 1 minute at the conclusion of the care episode.
- Total: Total of all reporting groups
Arm/Group | Experimental: Nurse-Administered Touch Intervention, Then Standard Care | Experimental: Standard Care, Then Nurse-Administered Touch Intervention | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 9 | 19
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: weeks gestation at birth] | 28.9 [27.3 to 30.7] | 28.7 [27.1 to 30.4] | 28.8 [27.1 to 30.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 9 | 6 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 19
Birthweight [Mean (Full Range); unit: grams] | 1339 [920 to 1967] | 1158.4 [870 to 1510] | 1253.5 [870 to 1967]

OUTCOME MEASURES:

1. Primary Outcome: Average Heart Rate -- During Intervention
Description: heart rate in beats per minute will be measured using an external electrocardiogram monitor and averaged over the intervention or control period
Time Frame: during intervention or control period, approximately 20 minutes
Population: 19 enrolled infants in randomized cross-over trial
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Nurse-Administered Touch Intervention | Standard Care
Number analyzed (Participants) | 16 | 16
beats per minute | 172.6 (10.5) | 168.6 (9.2)

2. Primary Outcome: Average Heart Rate -- Recovery
Description: as for outcome 1
Time Frame: recovery, 30 minutes after intervention delivery or control period
Population: 19 total infants participated in randomized cross-over trial
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Nurse-Administered Touch Intervention | Standard Care
Number analyzed (Participants) | 16 | 16
beats per minute | 161.7 (10.0) | 158.6 (8.4)

3. Secondary Outcome: Average High-frequency Heart Rate Variability -- During Caregiving Episode
Description: Spectral analysis of high-frequency heart rate variability averaged over the episode of caregiving during which infants received either the nurse-administered touch intervention or standard care. Spectral analysis of the high frequency band is a non-linear measure of heart rate variability that quantifies, primarily, parasympathetic nervous system (vagal) tone.
Time Frame: during caregiving episode that included either the nurse-administered touch intervention or was delivered as standard care, approximately 20 minutes
Population: 19 total participants in randomized cross-over trial
Measure: Median (Full Range); unit: ln(ms^2)
Arm/Group | Nurse-Administered Touch Intervention | Standard Care
Number analyzed (Participants) | 16 | 16
ln(ms^2) | 3.2 [2.1 to 4.8] | 3.2 [2.5 to 4.3]

4. Secondary Outcome: Average High-frequency Heart Rate Variability -- Recovery
Description: Spectral analysis of high-frequency heart rate variability averaged over the 30-minute period following caregiving that included the nurse-administered touch intervention or was delivered as standard care. Spectral analysis of the high frequency band is a non-linear measure of heart rate variability that quantifies, primarily, parasympathetic nervous system (vagal) tone.
Time Frame: recovery, 30 minutes after caregiving that included either the nurse-administered touch intervention or standard care
Population: 19 total participants in randomized cross-over trial
Measure: Median (Full Range); unit: ln(ms^2)
Arm/Group | Nurse-Administered Touch Intervention | Standard Care
Number analyzed (Participants) | 16 | 16
ln(ms^2) | 3.0 [2.1 to 5.5] | 3.0 [2.3 to 4.9]

5. Secondary Outcome: Average Frequency of Skin Conductance Responses -- During Caregiving Episode
Description: Frequency of skin conductance responses will be measured using an external monitor with electrodes attached to the infant's foot and averaged over the caregiving episode that includes either the nurse-administered touch intervention or standard care. Frequency is measured as number of waves per second over the duration of caregiving.
Time Frame: during caregiving episode, approximately 20 minutes
Population: 19 total participants in randomized cross-over trial
Measure: Mean (Standard Deviation); unit: waves per second
Arm/Group | Nurse-Administered Touch Intervention | Standard Care
Number analyzed (Participants) | 17 | 17
waves per second | 0.14 (0.05) | 0.14 (0.05)

6. Secondary Outcome: Average Frequency of Skin Conductance Responses -- Recovery
Description: Frequency of skin conductance responses will be measured using an external monitor with electrodes attached to the infant's foot and averaged over the 30-minute period following the caregiving episode that included either the nurse-administered touch intervention or standard care. Frequency is measured as number of waves per second over the duration of the 30-minute recovery period.
Time Frame: recovery, 30 minutes after intervention delivery or control period
Population: 19 total participants in randomized cross-over trial
Measure: Mean (Standard Deviation); unit: waves per second
Arm/Group | Nurse-Administered Touch Intervention | Standard Care
Number analyzed (Participants) | 17 | 16
waves per second | 0.06 (0.04) | 0.06 (0.05)

ADVERSE EVENTS:
Time Frame: Essential nursing care is scheduled to occur every 3 hours in the NICU. Study electrodes were attached to enrolled infants during the caregiving episode preceding the observed caregiving episode during which data collection occurred. Adverse events were documented from the time study electrodes were attached to the infant until the end of the 30-minute recovery period following the observed caregiving episode. Thus, total recording of adverse events was approximately 3.5 hours.
Description: standard definition applied
Arm/Group | Nurse-Administered Touch Intervention | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 5/19 | 8/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nurse-Administered Touch Intervention (N=19) | Standard Care (N=18)
bradycardia or oxygen desaturation (General disorders) | 5 (6) | 8 (8) — episode of bradycardia with heart rate <100 beats per minute for 10 seconds and/or oxygen desaturation with SpO2 <85% for 10 seconds

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT05030233/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT05030233/ICF_001.pdf